CLINICAL TRIAL: NCT01370018
Title: Zemaira (Alpha-1-Proteinase Inhibitor) Therapy in HIV-1 Disease
Brief Title: Therapy to Elevate CD4 Counts in HIV-1 Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institute for Human Genetics and Biochemistry (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Principal Investigator, Cynthia L Bristow, PhD, Assistant Professor, Mount Sinai School of Medicine, Institute for Human Genetics and Biochemistry
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R06-005
Record Dates: First submitted 2011-06-06; First posted 2011-06-09 (Estimated); Results first posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-08

CONDITIONS: HIV Disease
Keywords: CD4 counts; cholesterol
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — alpha 1-Antitrypsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- alpha-1 proteinase inhibitor in HIV (Experimental): HIV-1 infected individuals treated with Alpha-1 proteinase inhibitor
  Interventions: Biological: alpha-1-Proteinase Inhibitor

INTERVENTIONS:
Biological: alpha-1-Proteinase Inhibitor — Alpha-1-Proteinase Inhibitor was delivered I.V. A patient weighing 150 pounds was infused with approximately ½ cup containing 8.4 grams of alpha-1-Proteinase Inhibitor. Patients were admitted to hospital for infusion. The I.V. infusion was approximately 1 teaspoon/minute. Patients received weekly infusions of alpha-1-Proteinase Inhibitor for 8-12 weeks. At the time of infusion, 40ml (3 Tablespoons) of blood was collected (IRB approval #R04-003). The blood sample was used to monitor viral load, CD4 cell numbers, and alpha-1-Proteinase Inhibitor.
  Other Names: Zemaira; Prolastin

SUMMARY:
For more than 20 years, alpha-1-proteinase inhibitor therapy has been the standard treatment for patients who have inherited alpha-1-proteinase inhibitor deficiency. Adult patients with this condition eventually develop emphysema. Most HIV-1 patients who have low viral load also have alpha-1-proteinase inhibitor deficiency. The number of CD4 cells in blood increases when alpha-1-proteinase inhibitor increases. Patients will be asked to participate in a pilot study to see whether the use of Zemaira® (alpha-1-proteinase inhibitor) can increase blood levels of alpha-1-proteinase inhibitor and consequently increase CD4 counts.

DETAILED DESCRIPTION:
HIV-1 patients will be asked to participate in a pilot study to see whether the use of Zemaira increases blood levels of alpha-1-proteinase inhibitor and consequently increase CD4 counts.

HIV-1 patients will receive weekly treatment with Zemaira for 8 weeks by intravenous infusion. Blood will be collected immediately prior to each infusion. Blood will be collected at each visit. Exploratory assessments and not pre-specified outcome measurements will include complete blood count, lymphocyte phenotype, HIV-1 viral load, lipid levels, blood chemistry, and markers of inflammation from patient medical records. Exploratory and not pre-specified outcome measures will include extended lymphocyte phenotype and lymphocyte function using residual blood collected.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 patients must have confirmed HIV-1 disease, diagnosed using the standard criteria and be on antiretroviral therapy. Patients with inherited alpha-1 proteinase inhibitor deficiency (PIzz) must not have previously received alpha-1 proteinase inhibitor therapy. Uninfected volunteers will be age and gender matched.
2. HIV-1 patients must have measurable disease, defined as HIV-1 infected patients on antiretroviral therapy with undetectable HIV RNA (<500 HIV-1 RNA copies/ml) and CD4 counts more than 200 and less than 400 cells/uL.
3. Age at least 18 years and under 65 years.
4. HIV-1 patients must have active alpha-1 proteinase inhibitor below 11uM (normal is 18-53 uM).
5. HIV-1 patients must have one year history (prior to the study) with CD4 counts greater than 200 and less than 400 cells/uL.
6. Volunteers must have no evidence of malignancy.

Exclusion Criteria:

1. Recent illness that will prevent the patient from participating in required study activities.
2. Patients receiving other investigational agents.
3. Patients with known malignancies.
4. Patients with more than 500 HIV RNA copies/mL.
5. Patients with more than 400 CD4 cells/uL.
6. Uncontrolled illness including, but not limited to, ongoing or active infection, myeloid dysplastic syndrome, anemia, bone marrow failure, DiGeorge Syndrome, thymic disorders, or psychiatric illness/social situations that would limit compliance with study requirements.

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female subjects were not included in this pilot study to avoid pregnancy-related issues.
Enrollment: 4 (Actual)
Dates: Start 2006-12; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia L Bristow, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Jose Cortes, MD, Study Director — Beth Israel Medical Center
Locations (1):
- Cabrini Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bristow, C.L., Cortes, J., Mukhtarzad R., Trucy, M., Franklin, A., Romberg, V., Winston, R. 2010. α1Antitrypsin therapy increases CD4+ lymphocytes to normal values in HIV-1 patients. In Soluble Factors Mediating Innate Immune Responses to HIV Infection, (ed. M. Alfano). Bentham Science Publishers, http://www.alpha1biologics.com/BristowChapter.pdf
- [Result] Bristow CL, Modarresi R, Babayeva MA, LaBrunda M, Mukhtarzad R, Trucy M, Franklin A, Reeves RE, Long A, Mullen MP, Cortes J, Winston R. A feedback regulatory pathway between LDL and alpha-1 proteinase inhibitor in chronic inflammation and infection. Discov Med. 2013 Nov;16(89):201-18. PMID 24229737
- [Result] Bristow CL, Ferrando-Martinez S, Ruiz-Mateos E, Leal M, Winston R. Development of Immature CD4+CD8+T Cells Into Mature CD4+ T Cells Requires Alpha-1 Antitrypsin as Observed by Treatment in HIV-1 Infected and Uninfected Controls. Front Cell Dev Biol. 2019 Nov 21;7:278. doi: 10.3389/fcell.2019.00278. eCollection 2019. PMID 31824943

RESULTS

PARTICIPANT FLOW:
Groups:
- Alpha-1-Proteinase Inhibitor/HIV: This pilot study was performed to examine the efficacy of alpha-1 proteinase inhibitor augmentation in HIV-1 infected patients undergoing research treatment to elevate alpha-1-proteinase inhibitor and thereby, CD4 helper immune cells.
Period: Overall Study
Arm/Group | Alpha-1-Proteinase Inhibitor/HIV
Started | 4
Completed | 3
Not Completed | 1
Not completed — Did not meet criteria for analysis | 1

BASELINE CHARACTERISTICS:
Population: HIV patients were receiving antiretroviral medication with adequate suppression of virus. No patients had previously received alpha-1 proteinase inhibitor treatment.
Groups:
- Alpha-1-Proteinase Inhibitor in HIV: This pilot study was performed to examine the efficacy of alpha-1 proteinase inhibitor augmentation in 4 HIV-1 infected patients undergoing research treatment to elevate alpha-1-proteinase inhibitor and thereby, CD4 helper immune cells.Study subjects were evaluated at Baseline and weekly for at least 8 weeks.
Arm/Group | Alpha-1-Proteinase Inhibitor in HIV
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Sex/Gender, Customized [Number; unit: participants]
  Male | 4
  Female | 0
Region of Enrollment [Number; unit: participants]
  United States | 4
CD4 counts [Mean (Standard Deviation); unit: cells/uL] | 294 (125)
CD8 [Mean (Standard Deviation); unit: cells/uL] | 829 (281)
CD4/CD8 Ratio [Mean (Standard Deviation); unit: Ratio] | 0.40 (0.19)
active alpha-1 proteinase inhibitor [Mean (Standard Deviation); unit: μM] | 8 (3)

OUTCOME MEASURES:

1. Primary Outcome: CD4/CD8 Ratio
Time Frame: 9 weeks after initiation of treatment
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- Alpha-1-Proteinase Inhibitor in HIV: This pilot study was performed to show that Zemaira® treatment can be used in HIV-1 patients to elevate alpha-1-Proteinase Inhibitor and has the added benefit of elevating CD4 cells.
Arm/Group | Alpha-1-Proteinase Inhibitor in HIV
Number analyzed (Participants) | 3
Ratio | 0.44 (0.30)

ADVERSE EVENTS:
Time Frame: 9 weeks to 1 year post therapy
Groups:
- Alpha-1-Proteinase Inhibitor: This pilot study was performed to show that Zemaira® treatment can be used in HIV-1 patients to elevate alpha-1-Proteinase Inhibitor and has the added benefit of elevating CD4 cells.
Arm/Group | Alpha-1-Proteinase Inhibitor
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
One HIV infected patient enrolled, but entered the study with elevated inflammatory markers which were were not within the eligibility criteria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No